CLINICAL TRIAL: NCT01530516
Title: 3D Changes Comparing the Crossbow Appliance and Later Full Fixed Brackets Against Simultaneous Use of Full Fixed Brackets Plus Forsus Springs Among Mild to Moderate Class II Malocclusion Cases: A Randomized Clinical Trial.
Brief Title: Crossbow Versus Forsus Springs in Mild to Moderate Class II Malocclusion Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00021423
Record Dates: First submitted 2012-02-07; First posted 2012-02-10 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Malocclusion, Angle Class II
Keywords: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full brackets plus Forsus springs (Active Comparator): Standard of care - Class II springs used after le el and alignment.
  Interventions: Device: Brackets plus Forsus springs
- Xbow plus full brackets (Experimental): Alternative treatment - First use the Xbow appliance and then full brackets after Class II occlusion has been corrected.
  Interventions: Device: Xbow plus full brackets

INTERVENTIONS:
Device: Brackets plus Forsus springs — Full brackets and after completion of level and alignment insertion of Class II correctors (Forsus spring devices).
  Other Names: Forsus™ Fatigue Resistant Device
  Arms: Full brackets plus Forsus springs
Device: Xbow plus full brackets — Xbow appliance to be inserted first. After anteroposterior changes have been completed full brackets will be bonded and occlusion fine tuned
  Other Names: Xbow Class II corrector
  Arms: Xbow plus full brackets

SUMMARY:
Class II malocclusion (mismatch between the upper and lower jaw in which the lower jaw appears to be smaller from a profile point of view) are common in the general population. Around 1/3 of the population have some degree of this skeletal/dental problem and it is one frequent reason why patients decide to undergo orthodontic treatment. Treatment alternatives will basically depend on the facial skeletal development of the patient and also on the magnitude of the skeletal/dental discrepancy.

For patients that are not yet fully skeletal mature, the treatment of mild to moderate Class II malocclusion involves a combination of a small skeletal growth modification effect and more significant dental movements. For skeletal mature individuals with a severe mismatch, the treatment usually involves jaw surgery to fully correct the malocclusion. For less severe cases orthodontic camouflage exclusively done by orthodontic movements is an option.

If the case is not severe enough to warrant a surgical approach there are several treatment alternatives. One of the most commonly used options is the use of orthodontic loaded springs that apply forces through brackets and arch wires bonded into the teeth so that the teeth will interrelate better.

A different alternative was proposed some years ago. The Xbow (spelled Crossbow) appliance differs from the above-proposed option in that no brackets are bonded or arch wires used. The orthodontic springs are applied to a metal framework cemented on some upper and lower teeth. Once the skeletal/dental problem is believed to have been significantly improved, fine tuning of the remaining dental problems is managed with brackets and arch wires. The theoretical advantage of such a design is that adverse effects, such as root resorption and decalcification from the long-term use of brackets and arch wires, are theoretically minimized as the brackets and arch wires have to be used for a shorter period of time.

Although there are some retrospective reports about the skeletal and dental effects of the Xbow appliance and only one prospective trial comparing the skeletal and dental changes to a non-treated growing sample; no randomized clinical trial has yet evaluated the changes compared to a current standard of care alternative which is the simultaneous use of loaded springs concurrent with brackets and arch wires.

DETAILED DESCRIPTION:
Background

Class II malocclusion is a common orthodontic problem that requires comprehensive treatment planning. Treatment of Class II malocclusion is frequently initiated in mid to late mixed dentition whereby crowding and/or an increased over jet becomes alarming to patients and parents. Earlier correction of Class II abnormalities could be suggested in patients with significant occlusion discrepancies, increased risk of trauma to protruding upper incisors and impairment of mastication functions.

Among the available Class II correctors, cemented/fixed options are gaining popularity. Systematic reviews have shed some light on what fixed Class II correction devices appear to produce during treatment of mild to moderate Class II malocclusion. Short-term changes were a combination of skeletal and dental modifications. Skeletal modifications include both maxillary restriction and mandibular repositioning, and dental effects usually consist of inclination of mandibular incisors and maxillary molar distal movement.

Cephalometric analysis is a valuable tool used for diagnosis and treatment planning for dental malocclusion and underlying skeletal discrepancies. In view of the fact that a malocclusion is a product of an interaction between the alignment of the erupting teeth in their basal bone and the skeletal position of the basal bone itself, cephalometric analysis are used to evaluate dentoalveolar proportions and elucidate the anatomic basis for both jaw and tooth related abnormalities in the sagittal plane.

The Xbow appliance is a recently introduced orthodontic device that is used in late mixed or early permanent dentition before full fixed orthodontic treatment is initiated. Its main goal is to rapidly correct/improve the occlusion in a Class II malocclusion in mild to moderate cases. Full brackets thereafter will fine-tune the final occlusion.

Since its introduction there have been only three published studies of the Xbow appliance. One study focused on the evaluation of short-term skeletal and dental effects from lateral cephalograms while another discussed lower incisor inclination according to vertical facial types. Both reported mandibular incisor inclination of variable magnitude. The last published study analyzed if any conventionally utilized cephalometric variable was able to predict the amount of lower incisor inclination consistently.

As mentioned above, although the are some retrospective reports about the skeletal and dental effects of the Xbow appliance and only one pilot prospective trial comparing the skeletal and dental changes to a non-treated growing sample; no randomized clinical trial has yet evaluated the changes compared to a current standard of care alternative which is the simultaneous use of loaded springs concurrent with brackets and arch wires.

Objectives

The present study compares 3D facial, skeletal and dental changes using two orthopedic orthodontic approaches. Group 1 (alternative treatment) will use a fixed Class II corrector - Crossbow appliance - with full braces utilized later against Group 2 (one of the current available conventional treatments) with full fixed appliances with an additional fixed Class II corrector - (standard of care) - in clinical patients with mild to moderate Class II division 1 malocclusion.

An additional objective is to compare the adverse effects (root resorption and enamel decalcification) among both groups.

Methods

Each patient will undergo orthodontic clinical screening to determine if they fill the inclusion criteria (mild to moderate Class II malocclusion in a growing individual). Eligible candidates will be approached with an opportunity to participate in the research study. After understanding the research purpose and possible side effects, and they choose to participate, they will voluntarily sign the informed consent form. They will be randomly assigned to one of two groups. The researchers will not participate in the randomization as it would be done by a statistician and only communicated by phone once a participant is deemed to have fulfilled the inclusion criteria and provided informed consent.

Both treatment arms will start as soon as the randomization has been done. Full orthodontic records (digital volumetric images - Cone Beam Computer Tomograms, photos and dental casts) will be obtained for both groups at baseline and after treatment is completed.

Group 1 treatment will consist of fixed orthodontic appliances (brackets and molar tubes) with the addition of the spring loaded orthodontic corrector once occlusion level and alignment has been completed as per standard of care. It is expected that the treatment will last around 24 months.

Group 2 treatment will consist of a fixed functional Crossbow appliance. Bands will be fitted in the lower first molars, as well as in the upper first molars. A lingual and a vestibular arch connecting the lower molar bands, as well as a Hyrax type rapid maxillary expansion connecting the upper bands will be made in the laboratory. A Forsus spring will be connected from a molar tube in the upper first molar to lower vestibular arch with adjustable Guerin locks. It is expected that the Xbow treatment will be around 6 to 8 months. Fixed orthodontic appliances (brackets and molar tubes) will be inserted thereafter and the regular orthodontic treatment will be provided with an expected additional completion time of 12 to 16 months. Therefore total treatment time will be in the 24-month range.

A sample of 50 patients (25 patients per treatment group, considering a 20% loss during follow-up so that the groups will not have less than 21 patients per group at the end of study) will be sought. Assumptions made were with a SD of 5 degrees of lower incisor inclination, as averaged from previous studies, and a clinically significant difference of also 5 degrees.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be of either gender between 11 and 15 years-of-age.
* They will have mild to moderate Class II division 1 malocclusions.
* Late mixed dentition or early permanent dentition.

Exclusion Criteria:

* Severe vertical growth tendency or syndromic cases.
* Craniofacial growth completed.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Facial soft tissue, dental and skeletal changes | 24 months
  Outcomes to be measured from Computer Beam Computer Tomography data and dental casts.

SECONDARY OUTCOMES:
Root resorption | 24 months
  Evaluation of the magnitude of external root resorption as quantified/qualified from the CBCT data.
Enamel decalcification | 24 months
  Enamel decalcification as clinically determined by observing and touching the enamel surfaces of teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Flores Mir, DDS, FRCD(O), Principal Investigator — University of Alberta
Locations (1):
- Edmonton Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No